CLINICAL TRIAL: NCT02697942
Title: Hemodialysis-based Interventions to Preserve Cognitive Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: closure of dialysis center where study was being conducted
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00006466
Record Dates: First submitted 2016-02-09; First posted 2016-03-03 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Cognitive Training; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard of care (No Intervention): Participants randomized to the standard of care arm will not receive any intervention.
- Cognitive training (CT) (Experimental): Participants randomized to the CT arm will be given a tablet with connection to Lumosity®, which is a web-based "brain game". Participants will use the tablets to play brain games at each dialysis session.
  Interventions: Other: cognitive training
- Exercise training (ET) (Active Comparator): Participants randomized to ET arm will be given a stationary foot peddler. This foot peddler will be situated at a comfortable distance from the dialysis chair so that the patient can comfortably reach the peddler. Participants will use the foot peddlers at each dialysis session.
  Interventions: Other: exercise training

INTERVENTIONS:
Other: cognitive training — The investigators will provide participants with tablets to play brain games through Lumosity.
  Arms: Cognitive training (CT)
Other: exercise training — The investigators will provide participants with foot peddlers.
  Arms: Exercise training (ET)

SUMMARY:
This will be a pilot, single center, randomized, controlled trial to slow cognitive decline in adults undergoing hemodialysis (HD). The investigators will test two interventions (cognitive training and exercise training) against the standard of care.

DETAILED DESCRIPTION:
This will be a pilot, single center, randomized, controlled trial to slow cognitive decline in adults undergoing hemodialysis (HD). The investigators primary objective is to demonstrate feasibility for the interventions (cognitive training and exercise training) in Aim 1. The investigators will formally test whether whether cognitive training (tablet-based brain games) and exercise training (stationary foot pedal) administered during HD slow cognitive decline as well as improve secondary outcomes (physical function, frailty, and health-related quality of life (HRQOL) as part of Aim 2. The investigators will compare these two interventions against the standard of care. Pre- and post-intervention assessments will be conducted at the dialysis unit by a study coordinator and by research assistants. Participants will be followed for 6 months to assess cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with end stage renal disease and receiving hemodialysis at the DaVita Dialysis Centers located at 409 N. Caroline St., Baltimore, MD will be approached by our study coordinator to determine eligibility.

  * Must be at least 18 years or older at enrollment
  * Must be English speaking
  * Must be willing to participate in research and able to give informed consent

Exclusion Criteria:

* Chronic lung disease requiring oxygen
* Cerebrovascular disease
* Musculoskeletal conditions that limit mobility
* Lower or upper extremity amputation
* Orthopedic disorders exacerbated by physical activity
* Decreased mental capacity
* Dementia (diagnosed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Cognitive function measured using the Modified Mini Mental Status | 6 months post-intervention
  Cognitive decline assessed as both the change in Modified Mini Mental Status and Trail making Test A and B scores as well as 10% decline in these measures of cognitive function

SECONDARY OUTCOMES:
physical function measured using the Short Physical Performance Battery (SPBB) | 6 months post-intervention
  SPBB score of <10 considered as physical function impaired
Fried frailty phenotype | 6 months post-intervention
  Defined by the presence of 3 or more of the following: slowed walking speed, low physical activity, exhaustion, poor grip strength, and low physical activity. This is a binary outcome
health-related quality of life (HRQOL) | 6 months post-intervention
  measured by the Kidney Disease Quality of Life Scale
Cognitive function | 6 months post-intervention
  measured using the Trails Making Test A and B

CONTACTS AND LOCATIONS:
Overall Officials: Mara McAdams DeMarco, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Bond St DaVita Dialysis Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639